CLINICAL TRIAL: NCT06434038
Title: Measurement of Insulin Levels in the Cerebrospinal Fluid (CSF) of Healthy Adults After a Single Intranasal Dose - Middle Age
Brief Title: Measurement of Insulin Levels in the Cerebrospinal Fluid of Healthy Adults After a Single Intranasal Dose - Middle Age
Acronym: INI-CSF-MA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We are closing this clinical protocol due to supply chain issues. We are no longer able to obtain the intranasal delivery device.
Sponsor: HealthPartners Institute (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Department of Defense Congressionally Directed Medical Research Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A22-210; CDMRP-SC220220 (Other: Department of Defense)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: insulin; intranasal; Healthy Adults; Middle Age
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of 3 groups: 40 IU insulin, 80 IU insulin, or saline control.
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose intranasal insulin (Experimental): One dose of 40 international units of regular insulin administered intranasally.
  Interventions: Drug: Low Dose Regular insulin
- High dose Intranasal Insulin (Experimental): One dose of 80 international units of regular insulin administered intranasally.
  Interventions: Drug: High Dose Regular insulin
- Placebo Control (Placebo Comparator): One dose of 0.9% saline administered intranasally.
  Interventions: Other: 0.9% Saline

INTERVENTIONS:
Drug: Low Dose Regular insulin — Administered intranasally at 40 IU
  Other Names: Novolin-R
  Arms: Low dose intranasal insulin
Drug: High Dose Regular insulin — Administered Intranasally at 80 IU
  Other Names: Novolin-R
  Arms: High dose Intranasal Insulin
Other: 0.9% Saline — Placebo control
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to find out whether insulin, a drug approved by the FDA for the treatment of diabetes mellitus, reaches the brain and spinal cord when delivered as a nasal spray (intranasally). Intranasal insulin has been shown to improve memory and mood in patients with neurological diseases such as mild cognitive impairment and dementia, but more evidence is needed to support the ability to effectively target the brain through intranasal routes.

18 healthy middle-aged adults will be randomly assigned to receive a single intranasal dose of 40 units insulin ("low dose" group), 80 units insulin ("high dose" group), or saline (placebo, or control group). Participants will undergo an image-guided lumbar puncture (spinal tap) performed by a study clinician. Samples of cerebrospinal fluid (a fluid surrounding the brain and spinal cord) and blood will be collected at 5 timepoints during the lumbar puncture: once prior to the administration of intranasal insulin, and again at 10, 20, 30, and 40 minutes after the dose is given. Samples will be tested to determine the level of insulin detected in the cerebrospinal fluid and blood at each time point. Results of this study will provide essential information about the ability of insulin to reach the brain after intranasal administration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between ≥36 and ≤ 55 years of age
2. Subject's BMI is between >=18.5 and <=24.9, or can safely undergo a lumbar puncture at the discretion of the radiologist
3. MOCA score ≥26
4. Subject must be proficient in speaking English to comply with instructions and measures for the study
5. Subject can provide written informed consent
6. Female subjects must have either: (1) a negative pregnancy test at the screening visit and treatment visit OR (2) be at least 2 years post-menopausal / surgically sterile.

Exclusion Criteria:

1. Subject has medical history and/or clinically determined disorders: chronic sinusitis, previous nasal and/or oto-pharyngeal surgery and severe deviated septum and/or other anomalies.
2. Subject has history of any of the following: active and significant central nervous system, psychiatric illness, pulmonary, or cardiovascular disorders or any other clinically relevant abnormality that inclusion would pose a safety risk to the subject as determined by investigator
3. Subject has participated in a clinical trial investigation within 3 months of this study.
4. Subject has an insulin allergy
5. Subject has Insulin-dependent diabetes
6. Subject is pregnant or breast feeding
7. Contraindication to spinal tap or other safety factors that preclude lumbar puncture in the investigator's opinion
8. Any other clinically relevant finding that would pose a safety risk to the subject as determined by the investigator

Ages: 36 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Concentration of insulin over Time - Cerebrospinal fluid | 0-40 minutes post-intranasal administration
  Insulin concentration detected in cerebrospinal fluid at 5 time points (pre-insulin dose; and 10, 20, 30, 40 minutes after dose). Values will be reported as μIU/mL. Higher values indicate a greater concentration of insulin in the cerebrospinal fluid. Concentrations for each time point (overall and by dose) will be reported as a mean +/- standard error.
Cmax of insulin concentration- Cerebrospinal Fluid | 0-40 minutes post- intranasal administration
  CSF insulin concentration will also be reported by Cmax (peak concentration)
Tmax of insulin concentration-Cerebrospinal FLuid | 0-40 minutes post-intranasal administration
  CSF insulin concentration will also be reported by Tmax (time of peak concentration)
AUC (area under the curve) of insulin concentration-Cerebrospinal Fluid | 0-40 minutes post-intranasal administration
  CSF insulin concentration will also be reported by AUC (area under the curve, measured as time x concentration)

SECONDARY OUTCOMES:
Insulin Concentration Over Time- Serum | 0-40 minutes post-intranasal administration
  Insulin concentration detected in blood at 5 time points (pre-insulin dose; and 10, 20, 30, 40 minutes after dose). Values will be reported at μIU/mL. Higher values indicate a greater concentration of insulin in the blood. Concentrations for each time point (overall and by dose) will be reported as a mean +/- standard error.
Cmax of insulin concentration - Serum | 0-40 minutes post-intranasal adminitration
  Serum insulin concentration will also be reported by Cmax (peak concentration)
Tmax of insulin - Serum | 0-40 minutes post-intranasal administration
  Serum insulin concentration will also be reported by Tmax (time to peak concentration)
AUC (area under the curve) of insulin concentration - Serum | 0-40 minutes post-intranasal administration
  Serum insulin concentration will also be reported by AUC (area under the curve, measured as time x concentration).

CONTACTS AND LOCATIONS:
Overall Officials: Leah R Hanson, PhD, Principal Investigator — HealthPartners Institute; Kimberly Byrnes, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No